CLINICAL TRIAL: NCT05937100
Title: Clinical and Radiographic Evaluation of Hyaluronic Acid and Biodentine as Vital Pulpotomy Medications in Primary Molars: Randomized Controlled Clinical Trial
Brief Title: New Vital Pulpotomy Medications in Primary Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Weaam ibrahiem eltantawy, assistant lecturer at pediatric department-Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0103023PP
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Carious Exposure of Pulp
Keywords: Hyaluronic Acid - Biodentine - Pulpotomy
MeSH Terms: interventions — formocresol; tricalcium silicate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: the observer and the recipients will be blinded to the study group to avoid bias (double blind randomized controlled trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control: Formocresol (Active Comparator): Teeth will be treated by using squeezed sterile cotton pellet with 20% formcresol for 1 minute then removed and pulp stumps will be dressed with a layer of zinc oxide-eugenol (ZOE) paste.
  Interventions: Drug: Formocresol
- Group A : (Biodentine) (Experimental): The biodentine mix will be prepared according to the manufacturer's instructions and condensed lightly with a condenser on the pulp stumps, and allowed to set.
  Interventions: Drug: Biodentine
- Group B : (Hyaluronic acid gel) (Experimental): Hyaluronic acid gel will be compressed against the amputated pulp for 5 minutes. Then the pulp stumps will be dressed with a layer of zinc oxide-eugenol (ZOE) paste.
  Interventions: Drug: Hyaluronic acid gel

INTERVENTIONS:
Drug: Formocresol — Molars will be anesthetized by local anesthesia. The rubber dam will be used for isolation. Caries will be removed by large spoon excavator. When pulpal exposure occurs, deroofing of the pulp chamber will be achieved then pulpal tissue will be amputated using sharp excavator. Hemostasis will be obtained by applying pressure with saline moist cotton pellet. If bleeding has not stopped within 5 min, tooth will be excluded from the study.Teeth will be treated by using squeezed sterile cotton pellet with 20% formcresol for 1 minute
  Arms: control: Formocresol
Drug: Biodentine — Molars will be anesthetized by local anesthesia. The rubber dam will be used for isolation. Caries will be removed by large spoon excavator. When pulpal exposure occurs, deroofing of the pulp chamber will be achieved then pulpal tissue will be amputated using sharp excavator. Hemostasis will be obtained by applying pressure with saline moist cotton pellet. If bleeding has not stopped within 5 min, tooth will be excluded from the study.The biodentine mix will be prepared according to the manufacturer's instructions and condensed lightly with a condenser on the pulp stumps
  Arms: Group A : (Biodentine)
Drug: Hyaluronic acid gel — Molars will be anesthetized by local anesthesia. The rubber dam will be used for isolation. Caries will be removed by large spoon excavator. When pulpal exposure occurs, deroofing of the pulp chamber will be achieved then pulpal tissue will be amputated using sharp excavator. Hemostasis will be obtained by applying pressure with saline moist cotton pellet. If bleeding has not stopped within 5 min, tooth will be excluded from the study.Hyaluronic acid gel will be compressed against the amputated pulp for 5 minutes.
  Arms: Group B : (Hyaluronic acid gel)

SUMMARY:
Evaluate clinically and radiographically the effect of biodentine and hyaluronic acid (HA) versus formocresol (FC) as pulpotomy medications in primary molars.

DETAILED DESCRIPTION:
Split mouth randomized controlled clinical trial. This study will be conducted on 96 teeth from 48 children in age group 4-7 years and have bilateral lower primary molars indicated for vital pulpotomy procedure. for:

1. Clinical evaluation of biodentine, hyaluronic acid and formocresol groups according to presence of failure criteria at different follow up periods.
2. Radiographic evaluation of biodentine, hyaluronic acid and formocresol groups according to presence of failure criteria at different follow up periods.

ELIGIBILITY:
Inclusion Criteria:

* -Clinical criteria

  1. Restorable mandibular primary molars with deep carious lesions.
  2. Absence of gingival swelling or sinus tract.
  3. Absence of spontaneous pain
  4. Absence of pain on percussion. B-Radiographic Criteria: Absence of

  <!-- -->

  1. Discontinuity of lamina dura
  2. Internal root resorption.
  3. External root resorption.
  4. inter-radicular or periapical bone destruction (radiolucency)

Exclusion Criteria:

1. Excessive bleeding during pulp amputation.
2. Non vital/necrotic teeth.
3. Any sort of medical history contraindicating the pulp treatment.
4. Teeth approximate exfoliation
5. Patient's guardians are not intending to be part of the study.
6. Retreatment of previously pulpotomy treated molar -

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
clinically successful pulpotomy | 18 months
  1. Pain symptom - free teeth on percussion as well as during mastication.
  2. Absence of pathological tooth mobility.
  3. Absence of swelling of pulpal origin.
  4. . Absence of sinus tract.
radiographically successful pulpotomy | 18 months
  1. No internal or external root resorption.
  2. No periapical or furcation radiolucency.
  3. No widening of periodontal ligament space.

CONTACTS AND LOCATIONS:
Overall Officials: Weaam I El-tantawy, Principal Investigator — assistant lecturer ,Faculty of Dentistry, Mansoura University B.D.S (2016); Nadia M Farrag, Study Director — Professor ,Faculty of Dentistry, Mansoura University; Hossam E Hammouda, Study Director — Lecturer, Faculty of Dentistry, Mansoura University
Locations (1):
- Dentistry, Al Mansurah, Egypt